CLINICAL TRIAL: NCT02899923
Title: Register of Autoimmune Bullous Dermatoses
Acronym: REGIBUL
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO16091
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Autoimmune Bullous Dermatoses
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Autoimmune bullous dermatoses: Patients with autoimmune bullous dermatoses
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
Autoimmune bullous dermatoses are a group of diseases with chronic course. They are provoked by the production of autoantibodies against the dermal-epidermal junction or against the inter-keratinocyte junctions, resulting in the formation of intra-epidermal or sub-epidermal blisters.

The diagnosis of autoimmune bullous dermatoses is based on clinical and immunopathological findings, including skin direct immunofluorescence.

Systemic corticosteroid therapy is generally considered as the mainstay of treatment for many years both for bullous pemphigoid and pemphigus which are the most frequent diseases.

DETAILED DESCRIPTION:
The aim of the study is the creation of a register of patients suffering from autoimmune bullous dermatoses to quickly identify patients who can be included in clinical trials or retrospective epidemiological studies

ELIGIBILITY:
Inclusion Criteria:

* patients with autoimmune bullous dermatosis
* patients cared for in dermatology referral center of Reims, Rouen or Limoges
* patient consenting to participate to the study

Exclusion Criteria:

- patient <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autoimmune bullous dermatosis
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
autoimmune bullous dermatosis according to physical examination, skin biopsy and autoantibodies detection in blood sample | Day 0
  Each autoimmune bullous dermatosis is classified according one of the following diagnoses : 1/ bullous pemphigoid, 2/ Mucous membrane pemphigoid, 3/ Pemphigoid gestationis, 4/ Epidermolysis bullosa acquisita, 5/ Linear IgA bullous dermatosis, 6/ pemphigus (vulgaris or foliaceus)
  This classification will be performed according :
  * clinical characteristics including location, clinical aspect and number of cutaneous and/or mucosal blisters
  * skin biopsy for routine histology (subepidermal blister or intra-epidermal blister) and direct immunofluorescence (IgG and/or I gA and/or C3 deposits along the epidermal basement membrane zone or on the cell surface of keratinocytes)
  * blood sample for serum autoantibodies detection against epidermal autoantigens using ELISA or indirect immunofluorescence techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France